CLINICAL TRIAL: NCT00533806
Title: Family Based Treatment for Early Childhood OCD
Brief Title: Comparing the Effectiveness of Two Family-based Therapies in Treating Young Children With Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer B. Freeman, Director, Outpatient Child Psychiatry; Staff Psychologist, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH079217 (NIH); R01MH079217 (NIH); DSIR 84-CTS
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Cognitive Behavior Therapy; Active Control; Relaxation Therapy; Young Children
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive behavioral therapy (Experimental): Participants will receive cognitive behavioral therapy.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Relaxation therapy. (Active Comparator): Participants will receive relaxation therapy.
  Interventions: Behavioral: Relaxation Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — CBT includes 12 treatment sessions over 14 weeks. The sessions deliver family-based exposure with response prevention. Participants assigned to receive CBT will learn skills to help control OCD. CBT sessions will also include education about OCD, family therapy, parent training to manage child behavior problems, and anxiety management.
  Arms: Cognitive behavioral therapy
Behavioral: Relaxation Therapy — Relaxation therapy includes 12 sessions delivered over 14 weeks. Participants assigned to receive relaxation therapy will discuss general family functioning, issues related to OCD, and other behavioral problems the child may be experiencing.
  Arms: Relaxation therapy.

SUMMARY:
This study will compare the effectiveness of family-based cognitive behavioral therapy to family-based relaxation therapy in treating young children with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a type of anxiety disorder that affects approximately 1 in 200 children. Although feelings of anxiety, fear, and uncertainty are a normal part of life and growing up, for some children these feelings and emotions become chronic, relentless, and progressively worse if left untreated. OCD is characterized by obsessions, or repeated unsettling thoughts, causing a person to perform repeated actions called compulsions. Children are typically not diagnosed with OCD until they are between the ages of 8 and 12, leaving many young children undiagnosed. Additionally, no psychotherapy treatments have been designed for young children who are under the age of 8 and have OCD. The purpose of this study is to develop and evaluate a family-based treatment program for children, ages 5 to 8, who have been diagnosed with OCD.

Participants in this open-label study will be randomly assigned to receive either cognitive behavior therapy (CBT) or relaxation therapy for 12 sessions over a period of 14 weeks. All children will undergo a 3-hour screening that will include a psychiatric evaluation and the completion of questionnaires. Parents of participating children will attend the first two treatment sessions without their children during which they will be introduced to the treatment program and will learn various skills to be used throughout treatment. The other 10 1-hour sessions will be attended by both the parent and child. Participants assigned to receive CBT will learn skills to help control OCD. Education about OCD, family therapy, parent training to manage child behavior problems, and anxiety management will be included in the CBT sessions. Participants assigned to receive relaxation therapy will discuss general family functioning, issues related to OCD, and other behavioral problems the child may be experiencing. Treatment will also include education about OCD; affective education, during which participants will learn how to recognize feelings; muscle relaxation techniques; and guided imagery. Participants in both treatment groups will receive weekly homework assignments after each session to practice skills learned. Parents will also be asked to monitor their child's behavior and practice the learned skills with their child as often as possible. If treatment has not been successful after the 14-week period, the child will be offered an alternative treatment. All participants will be assessed before treatment; at 5, 9, and 14 weeks of treatment; and at 3, 6, and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for OCD
* Parent willing to sign informed consent

Exclusion Criteria:

* History or current diagnosis of pervasive developmental disorder(s), thought disorder, or mental retardation
* Psychotic symptoms

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale | Measured immediately post-treatment and at Months 3, 6, and 12

SECONDARY OUTCOMES:
Clinical Global Improvement | Measured immediately post-treatment and at Months 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B. Freeman, PhD, Principal Investigator — Rhode Island Hospital/ Brown Medical School; Marty Franklin, PhD, Principal Investigator — University of Pennsylvania; John S. March, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Child and Family Study Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown Medical School/ Rhode Island Hospital/ Pediatric Anxiety Research Clinic, Providence, Rhode Island

REFERENCES:
- [Derived] Freeman J, Sapyta J, Garcia A, Compton S, Khanna M, Flessner C, FitzGerald D, Mauro C, Dingfelder R, Benito K, Harrison J, Curry J, Foa E, March J, Moore P, Franklin M. Family-based treatment of early childhood obsessive-compulsive disorder: the Pediatric Obsessive-Compulsive Disorder Treatment Study for Young Children (POTS Jr)--a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):689-98. doi: 10.1001/jamapsychiatry.2014.170. PMID 24759852
- See also: Click here to visit the Obsessive Compulsive Foundation's Web site — http://www.ocfoundation.org